CLINICAL TRIAL: NCT07388173
Title: Assessment of Functional Impact of Acute Respiratory Viral Infections in Older Adults - An International Multi-center Study
Brief Title: Functional Impact of Acute Respiratory Viral Infections in Older Adults
Acronym: AFIRI
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC25.0367
Record Dates: First submitted 2025-12-29; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Infections in Old Age
Keywords: functional dependency; respiratory infection; elderly people
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevention of infectious diseases in older adults remains a major public health challenge, as acute respiratory infections are a leading cause of hospitalisation, mortality, and functional decline worldwide. Immunosenescence and environmental exposures increase susceptibility to infection and reduce vaccine effectiveness in this population. Respiratory viruses, including influenza, SARS-CoV-2, respiratory syncytial virus, and human metapneumovirus, account for a substantial share of this burden, much of which is vaccine-preventable. However, their impact on functional decline and recovery in older adults remains insufficiently characterized. This international study aims to assess the effect of hospitalization for major respiratory viral infections on loss of autonomy in individuals aged 60 years and older, to inform targeted prevention and vaccination strategies.

DETAILED DESCRIPTION:
The prevention of infectious diseases in older adults represents a major public health challenge due to their substantial impact on morbidity, mortality, and loss of functional capacity. Acute respiratory infections are among the leading causes of hospitalization and death in this population worldwide.

Ageing is associated with a progressive decline in immune function, resulting in increased susceptibility to infections and reduced vaccine effectiveness. In addition, environmental factors such as residence in collective living settings and repeated exposure to healthcare environments further increase the risk of exposure to and transmission of infectious agents.

The pathogens most frequently involved include respiratory viruses namely influenza, SARS-CoV-2, respiratory syncytial virus, and human metapneumovirus as well as bacterial pathogens, particularly Streptococcus pneumoniae, and certain fungal agents. A substantial proportion of these infections are potentially preventable through vaccination.

Despite advances generated by the European IMI VITAL project and the AEQUI case-control study, data remain limited regarding the functional consequences of acute respiratory infections in older adults, particularly their impact on dependency, frailty, and post-infectious recovery.

This international study aims to address these knowledge gaps by evaluating the impact of hospitalizations related to influenza, SARS-CoV-2, respiratory syncytial virus, and human metapneumovirus on loss of autonomy in individuals aged 60 years and older. The findings are expected to strengthen the scientific evidence base needed to inform targeted vaccination and prevention strategies, ultimately contributing to healthier ageing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 60 years or older
* Hospitalized in a study center (emergency department, infectious disease, internal medicine or geriatric hospital wards…) for acute respiratory infection (refer to table 1 below for definition).
* Confirmed positive PCR test for influenza, SARS-CoV-2, RSV, or human metapneumovirus (hMPV). Participants with co-infections with other viral or bacterial agents can be included.

Exclusion Criteria:

* Participants with conditions significantly impacting short-term functional status, such as severe disability (ADL score ≤2 or Clinical Frailty Scale ≥7), terminal illness, palliative care needs, or inability to comprehend and complete study questionnaires due to severe stroke sequelae, complete sensory loss, advanced dementia, or similar impairments.
* Participants that refuse or are unable to answer the 3- and 6-months follow-up phone call assessments
* Positive laboratory test for single (mono-infection) virus other than influenza, SARS-CoV-2, RSV, or human metapneumovirus (HMPV)
* Participant in exclusion period for another study using an investigational / unapproved medicinal product.
* Participant referred to in articles L1121-5 to L1121-8 of the CSP (corresponding to all protected persons : pregnant woman, parturient, breastfeeding mother, person deprived of liberty by judicial or administrative decision, persons undergoing psychiatric care under articles L.3212-1 and L.3213-1 who do not fall under article L.1121-8, persons admitted to a healthcare or social institution for purposes other than research, minors, person under legal protection or unable to express consent).
* Individuals opposed to participating in the research
* Staff members with a hierarchical relationship to the principal investigator

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will include participants aged 60 years or older who are hospitalized with a serious acute respiratory infection in the departments of infectious diseases, geriatrics, internal medicine, pulmonology, or emergency medicine. Recruitment will be conducted by investigator physicians in each participating department. Potentially eligible participants will be identified by daily screening of admission records and results from standard of care respiratory samples.
  Each country will aim to recruit approximately 320 participants - 80 with each pathogen of interest. Efforts will be made to secure an equal distribution of participants aged 60-75 and >75 years age.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Evolution of Functional Dependency assessed by Activities of Daily Living (ADL) Score | Baseline, at hospital discharge, 3 months after discharge, and 6 months after discharge.
  Change in functional performance measured using the Activities of Daily Living (ADL) scale. The ADL score ranges from 0 to 6, where higher scores indicate better functional independence The ADL score ranges from 0 to 6, where higher scores indicate better functional independence.
Evolution of Functional Dependency assessed by Instrumental Activities of Daily Living (IADL) Score | Baseline, Day 7, 3 months after discharge, and 6 months after discharge.
  Change in functional performance measured using the Instrumental Activities of Daily Living (IADL) scale. The IADL score ranges from 0 to 8, where higher scores indicate better functional independence.

SECONDARY OUTCOMES:
Functional Status depending on Viral Etiology Assessed by Activities of Daily Living (ADL) Score | Baseline, Day 7, 3 months after discharge, and 6 months after discharge.
  Change in functional status measured using the Activities of Daily Living (ADL) scale.
  The ADL score ranges from 0 to 6, where higher scores indicate better functional independence. Changes in score will be assessed between baseline, hospital discharge, 3 months, and 6 months, and stratified by viral etiology (SARS-CoV-2, influenza, respiratory syncytial virus (RSV), and human metapneumovirus (hMPV)).
Functional Status depending on Viral Etiology Assessed by Instrumental Activities of Daily Living (IADL) Score | Baseline, Day 7, 3 months after discharge, and 6 months after discharge.
  Change in functional status measured using the Instrumental Activities of Daily Living (IADL) scale. The IADL score ranges from 0 to 8, where higher scores indicate better functional independence.
  Changes in score will be assessed between baseline, hospital discharge, 3 months, and 6 months, and stratified by viral etiology (SARS-CoV-2, influenza, respiratory syncytial virus (RSV), and human metapneumovirus (hMPV)).
Medical Complications during and after hospitalization | From hospital admission to 6 months after discharge.
  Occurrence of medical complications during hospitalization and up to 6 months after discharge, including new diagnoses identified during follow-up.
Health Care Resource Utilization (HCRU) | From hospital admission to 6 months after discharge.
  Health care resource utilization, including hospital length of stay, intensive care unit (ICU) admission during index hospitalization, and hospital readmissions occurring between discharge and 6 months.
Length of Hospital Stay | 3 months after discharge
  Duration of the index hospitalization, measured in days, calculated from hospital admission (Day 1) to hospital discharge.
Intensive Care Unit (ICU) Admission | 3 months after hospital discharge.
  Proportion of participants admitted to an intensive care unit during the index hospitalization.
Hospital Readmissions After Discharge | From at hospital discharge to 6 months after discharge.
  Occurrence of hospital readmissions between discharge and 6 months after discharge.
New Medications Initiated | From hospital admission to 6 months after discharge.
  Initiation of new drug treatments during hospitalization or within 6 months after discharge.
Discharge Location after Hospitalization | 3 months after hospital discharge.
  Location at hospital discharge (e.g., home, rehabilitation facility, long-term care facility).
Living Situation at 6 Months after Discharge | 6 months after hospital discharge.
  Living situation of participants at 6 months after hospital discharge
Demographic Characteristics of Participants | Baseline.
  Baseline demographic characteristics of participants, including age and sex.
Living Situation at Baseline | Baseline.
  Living situation of participants prior to hospital admission.
Prevalence of Comorbidities | Baseline.
  Prevalence of pre-existing comorbidities at baseline.
Vaccination Status | Baseline.
  Proportion of participants vaccinated against influenza, SARS-CoV-2, and respiratory syncytial virus (RSV).
Time since last vaccination | Baseline.
  Time elapsed since the most recent vaccination against influenza, SARS-CoV-2, or RSV, measured in months.
Pneumonia Severity Index (PSI) Score | Baseline
  Severity of pneumonia assessed using the Pneumonia Severity Index (PSI) score at hospital admission.

CONTACTS AND LOCATIONS:
Locations (24):
- University of Rochester School of Medicine, Infectious Diseases Unit, Rochester, New York, United States
- France (6):
  - University Hospital of Amiens, Amiens
  - Melun Hospital, Melun
  - Villeneuve Saint Georges Hospital, Paris
  - University Hospital of Poitiers, Poitiers
  - University Hospital of Reims, Reims
  - University Hospital of Tours, Tours
- Germany (5):
  - Klinikum Bayreuth, Klinik für Geriatrie, Bayreuth
  - Abteilung Geriatrie Universitätsmedizin Göttingen, Abteilung Geriatrie, Göttingen
  - Uniklinikum Jena, Klinik für Geriatrie, Jena
  - Universitätsmedizin Mannheim, IV. Medizinische Klinik (Geriatrie), Mannheim
  - Klinikum Ulm, Geriatrisches Zentrum Agaplesion Bethesda, Ulm
- Italy (9):
  - University of Bari, Bari, Bari
  - Azienda Ospedaliero Universitaria "Renato Dulbecco", Catanzaro, Catanzaro
  - ULSS 5 Polesana, Rovigo, Rovigo
  - ASL 1 Imperiese, Sanremo, Sanremo
  - Città di Torino, Torino, Torino
  - APSS Trento, Geriatria, Trento, Trento
  - ASUGI, Trieste, Trieste
  - ULSS 3 Serenissima, Venice, Venice
  - ULSS 9 Scaligera, Legnago, Verona, Verona
- Spain (3):
  - Hospital Clínic Barcelona Servicio de Geriatría, Barcelona
  - Hospital Universitario Ramón y Cajal. Madrid Servicio de Geriatría, Madrid
  - Hospital Universitario Virgen de la Arrixaca Murcia Servicio de Geriatría, Murcia